CLINICAL TRIAL: NCT01010802
Title: Phase 1 Study of Recombinant Human Erythropoietin (rhEPO) in Parkinson's Disease (PD)
Brief Title: Safety Study of Erythropoietin (EPO) in Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Center for Neurological Restoration, Cuba (Other)
Collaborators: Centro de Immunologia Molecular, Cuba (Industry)
Responsible Party: Principal Investigator, Ivonne Pedroso Ibanez, Head of the Movement Disorders Clinic, International Center for Neurological Restoration, Cuba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EPO-001-PD
Record Dates: First submitted 2009-11-08; First posted 2009-11-10 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease
Keywords: Neuroprotection; Parkinson Disease; Erythropoietin
MeSH Terms: conditions — Parkinson Disease | interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erythropoietin (Experimental): There are evidences of neuroprotecting therapeutic alternatives in such substances as erythropoietin (EPO) which is a well-known cytokine as a hematopoietic growth factor, so, it is therefore important to control tissular oxygenation. It is considered that EPO protects the neurons by a combination of several mechanisms.
  EPOrh is used with high effectiveness in the treatment of anemias with deficiency of erythropoietin.
  Interventions: Drug: Erythropoietin human recombinant (EPOrh)

INTERVENTIONS:
Drug: Erythropoietin human recombinant (EPOrh) — Administration scheme by subcutaneous via, of an EPOrh solution up to a weekly doses of 60 UI/kg for five weeks
  Other Names: EPOCIM® (Center of Molecular Immunology, Habana, Cuba)

SUMMARY:
The purpose of this study is to determine whether recombinant human Erythropoietin (EPOrh) is safe in the treatment of patients with Parkinson's Disease.

DETAILED DESCRIPTION:
After onset of Parkinson's Disease (PD)- in spite of the use of medications that constitute the symptomatic treatment- the disease is worsens with an inevitable progression, thus causing complications that lead to the loss of patient´s manual skills and independent gait. At present, the treatment of PD with the use of medications is based on dopamine precursors and dopaminergic agonists but as the disease advances, other symptoms that do not respond to dopaminergic stimulation do appear.

For this reason, it is a priority to find a way to focus on neuroprotection during the course of the disease. There are evidences of neuroprotecting therapeutic alternatives in such substances as erythropoietin (EPO).

Positive results on the neuroprotective/neurotrophic efficacy of EPO in neurological and psychiatric diseases have been obtained from treatment trials, but nevertheless, it is indispensable demonstrate that with the proposed medication doses it's well tolerated by PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Hohen and Yahr´s Scale between I and III
* One or more years of evolution of PD,
* Good response to levodopa (more that 30 % of change)valued in motor UPDRS
* An acceptable general health status,

Exclusion Criteria:

* Chronic psychiatric or other neurological diseases.
* Previous polyglobulin
* Hematocryte, same or inferior to 50

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
safety assessment measured by the absence of adverse events | weeks 1 to 5, 6, 12, 23 and 35

SECONDARY OUTCOMES:
Post-treatment change in the motor score of the Unified Assessment Scale for Parkinson Disease´s (UPDRS) in the "OFF" condition as compared with the baseline. | week 6, 12, 23 and 35

CONTACTS AND LOCATIONS:
Overall Officials: Ivonne Pedroso, M.D., M.Sc., Principal Investigator — International Center for Neurological Restoration; Lazaro M Alvarez, M.D., Study Director — International Center for Neurological Restoration
Locations (1):
- Clinic of Movement Disorders, International Center for Neurological Restoration, Havana, Cuba

REFERENCES:
- [Result] Pedroso I, Bringas ML, Aguiar A, Morales L, Alvarez M, Valdes PA, Alvarez L. Use of Cuban recombinant human erythropoietin in Parkinson's disease treatment. MEDICC Rev. 2012 Jan;14(1):11-7. doi: 10.37757/MR2012V14.N1.4. PMID 22334107
- [Result] Pedroso I, Garcia M, Casabona E, Morales L, Bringas ML, Perez L, Rodriguez T, Sosa I, Ricardo Y, Padron A, Amaro D. Protective Activity of Erythropoyetine in the Cognition of Patients with Parkinson's Disease. Behav Sci (Basel). 2018 May 21;8(5):51. doi: 10.3390/bs8050051. eCollection 2018 May. PMID 29862060